CLINICAL TRIAL: NCT02489838
Title: Analysis of Lung Dose Using Volumetric Analysis in Patients Treated With Yttrium-90 Microsphere Radioembolization for Hepatocellular Carcinoma
Brief Title: Lung Dose in Patients Treated With Yttrium-90 for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Alan Katz (Other)
Responsible Party: Sponsor-Investigator, Alan Katz, Associate Professor, Radiation Oncology, University of Rochester
Organization: University of Rochester (Other)
Other Study IDs: ULAB11069
Record Dates: First submitted 2014-12-24; First posted 2015-07-03 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Liver Neoplasms
Keywords: Liver Neoplasma; Lung Radiation dose
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To Calculate the amount radiation the lung receives in patients receiving Yttrium-90 for Liver Cancer.

DETAILED DESCRIPTION:
To calculate the delivered lung dose using quantitative volumetric analysis in a cohort of patients with unresectable hepatocellular carcinoma who undergo selective internal radiation therapy (SIRT) with Yttrium-90 glass microspheres (TheraSphere®)-and compare this analysis to the lung dose estimated by established criteria. In addition, this study, will summarize the pre and post-treatment clinical data to describe the URMC Y-90 experience.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years with no upper limit.-Receiving Y-90 Therasphere liver directed therapy
* Pathology proven diagnosis of hepatocellular carcinoma, metastatic colon cancer or other metastatic diseases to be treated with SIRT (Y-90)
* surgical resection not feasible at time of initiation of pre-treatment workup

  -> 6 months projected life span
* ECOG 0-2

Exclusion Criteria:

* previous radioembolization of one or more liver lobes or segments without available treatment planning and procedural documentation ie. at another facility prior to URMC Y-90 radioembolization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Patients at the University of Rochester
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-02-03 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Lung dose measured with actual lung mass vs Lung dose measured with conventional method. | 1 month after treatment.
  Lung dose measured with actual lung mass vs Lung dose measured with conventional method which assumes 1 kg for all patients.
  Patient will be receiving this treatment even if not enrolled on this study.
  The study is NOT about the intervention given to the patient. The study is to determine the best way to measure the radiation dose normal tissue (the lung specifically) receives during this standard treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Katz, MD, Principal Investigator — Universtiy of Rochester
Locations (1):
- Radiation Oncology, University of Rochester, Medical Center, Rochester, New York, United States